CLINICAL TRIAL: NCT02742025
Title: Evaluation of the Effect of an Educational and Explanatory Program for a Surgical Act Provided to the Patient Prior to Said Act on Preoperative Anxiety - a Pilot Study at the Nîmes University Hospital on Elective Coronary Angiography
Brief Title: Effect of an Educational and Explanatory Program for a Surgical Act on Preoperative Anxiety
Acronym: HEART-LINK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: LOCAL/2016/EB-01
Record Dates: First submitted 2016-04-07; First posted 2016-04-18 (Estimated); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Preoperative Anxiety
Keywords: Coronary Angiography

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (Other): Patients randomized to this arm will have standard care with no extra interventions.
  Intervention: Inclusion visit
  Intervention: Coronarography on day 0
  Interventions: Other: Inclusion visit; Procedure: Coronarography on day 0
- HEARTLINK (Experimental): Patients randomized to this arm will participate in the HEARTLINK program, which includes a specific nurse consultation and telephone contact.
  Intervention: Inclusion visit
  Intervention: Nurse consultation
  Intervention: Telephone contact
  Intervention: Coronarography on day 0
  Interventions: Other: Inclusion visit; Other: Nurse consultation; Other: Telephone contact; Procedure: Coronarography on day 0

INTERVENTIONS:
Other: Inclusion visit — This visit takes place between days -15 and -7 preceding a coronarography scheduled for Day 0. It is part of standard care and corresponds to a required cardiology consultation.
Other: Nurse consultation — This visit takes place on the same day as the inclusion visit and includes practical advice concerning the hospital stay, explanations concerning the surgical act and practical advice on its implementation, information on the length of stay and after. An explanatory booklet concerning the surgical procedure is provided to the patient.
  Arms: HEARTLINK
Other: Telephone contact — A nurse will telephone the patient 72h to 48h before the coronarography scheduled for day 0. During the telephone conversation the nurse will assess the patient's knowledge about his/her pathology, his/her examination and the course of hospitalization. The nurse will answer any questions and if needed provide further information.
  Arms: HEARTLINK
Procedure: Coronarography on day 0 — This coronarography is scheduled as part of the patient's routine care. This is not an experimental intervention under evaluation.

SUMMARY:
The main objective of this study is to evaluate the impact on preoperative anxiety of an education and information program conducted prior to non-urgent coronary angiography performed in patients hospitalized at the Nîmes University Hospital.

DETAILED DESCRIPTION:
The secondary objectives of this study are to assess the impact of the HEARTLINK program on the following parameters:

A. Duration of hospital stay; B. Per operative blood and heart rate?; C. Patient satisfaction (visual analog scale).

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* Patient for whom elective coronary angiography is indicated
* The patient has never had a coronary angiography before

Exclusion Criteria:

* The patient is participating in another study
* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection, under tutorship or curatorship
* The patient refuses to sign the consent
* It is impossible to correctly inform the patient
* The patient is pregnant or breastfeeding
* The subject has already had a coronary angiography
* The subject has a cognitive impairment

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2019-11-19 (Actual); Primary Completion 2022-05-10 (Actual); Study Completion 2022-05-10 (Actual)

PRIMARY OUTCOMES:
Amsterdam Preoperative Anxiety and Information Scale (APAIS) | Day 0 (within 1 hour preceding a coronography)

SECONDARY OUTCOMES:
Duration of hospitalization | Date hospital discharge (expected maximum of 5 days)
Blood pressure | Day 0 (within 1 hour preceding a coronography)
Cardiac frequency (beats per minute) | Day 0 (within 1 hour preceding a coronography)
Visual analog scale for satisfaction concerning care | Day 0 (within 1 hour preceding a coronography)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Baljou, IDE, Study Director — Centre Hospitalier Universitaire de Nîmes
Locations (1):
- CHRU de Nîmes - Hôpital Universitaire Carémeau, Nîmes, France